CLINICAL TRIAL: NCT04424134
Title: Open Label Randomized Clinical Trial BromhexIne And Spironolactone For CoronаVirUs Infection Requiring HospiTalization
Brief Title: BromhexIne And Spironolactone For CoronаVirUs Infection Requiring HospiTalization
Acronym: BISCUIT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lomonosov Moscow State University Medical Research and Educational Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSU160520
Record Dates: First submitted 2020-05-27; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: COVID 19
Keywords: COVID 19; bromhexine; spironolactone
MeSH Terms: conditions — COVID-19 | interventions — Bromhexine; Spironolactone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bromhexine And Spironolactone (Experimental)
  Interventions: Drug: Bromhexine and Spironolactone
- Base therapy (Active Comparator)
  Interventions: Drug: Base therapy

INTERVENTIONS:
Drug: Bromhexine and Spironolactone — Bromhexine 8 mg x 4 times a day x 10 days Spironolactone 50 mg x once a day x 10 days
  Arms: Bromhexine And Spironolactone
Drug: Base therapy — Therapy currently recommended by Ministry of Health of Russian Federation for COVID 19 treatment
  Arms: Base therapy

SUMMARY:
Patients with mild and severe COVID 19 will be randomized 1:1 into two groups: experimental, which will get bromhexine and spironolactone, and control. Patients will get investigated therapy for ten days. Change in clinical assessment score COVID 19 (CAS COVID 19) between baseline and 12th day will be evaluated as a primary endpoint. Forty-five-day risk of death or mechanical ventilation will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

signed inform consent COVID 19 with the mild and severe course. The diagnosis could be made with positive polymerase chain reaction (PCR) (International Statistical Classification (ICD-10) code - U07.1) and/or virus pneumonia in computer tomography (ICD 10 code - U07.2) 5. Lung exposure on CT more than 25% 6. Sp02 without supportive oxygen ≤ 93% 7. C-reactive protein > 60 mg/l or elevation of C reactive protein 3 times in 8-14 days after first symptoms

Exclusion Criteria:

* pregnancy and breastfeeding
* hypersensitivity to Spironolactone
* hypersensitivity to Bromhexine
* Known liver failure
* Glomerular filtration rate <20 ml/ min
* physician judgment that the patient will need mechanical ventilation in 24 hours
* other indications for Spironolactone
* Active cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-05-16 (Actual); Primary Completion 2020-07-18 (Estimated); Study Completion 2020-08-23 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in clinical assessment score COVID 19 (CAS COVID 19) | baseline, day 12
  change in CAS COVID 19 between baseline and 12th +/- 2 days
  CAS COVID 19 measures clinical and laboratory parameters in 7 domains:
  respiratory rate (< 18 - 0 point; 18-22 - 1 point; 23-26 - 2 point; >26 - 3 point) body temperature (35.5 - 37.0 - 0 point; < 35.5 - 1 point; 37.1 - 38.5 - 1 point; > 38.5 - 2 point) Sp02 without support oxygen (> 93% - 0 point; 90-93% - 1 point; < 90% - 2 point) ventilation (not required - 0 point; low-flow ventilation - 1 point; Non-invasive positive pressure ventilation - 2 point; mechanical ventilation - 3 point) C-reactive protein (> 10 - 0 point; 10-59 - 1 point; 60-120 - 2 point; > 120 - 3 point) d - dimer (< 0.51 - 0 point; 0.51 - 2.0 - 1 point; 2.01 - 5.0 - 2, > 5.0 - 3 point) exposure area on lung CT (no pneumonia - 0; 1-24% - 1 point; 25-50% - 2; 51-75% - 3, > 75% - 4).
  Minimal number of points - 0; max - 20.Lower the score-better health

SECONDARY OUTCOMES:
- Combine endpoint - | 12 days, 45 days
  time to death or mechanical ventilation
C-reactive protein | 12 days, 45 days
  - Change from baseline in C-reactive protein
D-dimer | 12 days, 45 days
  - Change from baseline in D-dimer
EuroQol Group. EQ-5D™ | 12 days, 45 days
  Change from baseline in EQ-5D.
  The EQ-5D descriptive system comprises the 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box to the most appropriate statement. This decision results into a 1-digit number, . The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
EuroQol Group. EQ VAS | 12 days, 45 days
  Change from baseline in EQ VAS
  EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. The VAS can be used as a quantitative measure of health outcome by patient's own judgement.
HADS | 14 days, 45 days
  - Change from baseline Hospital Anxiety and Depression Scale/The Hospital Anxiety and Depression Scale (HADS) is a 14-item measure designed to assess anxiety and depression symptoms in medical patients, with emphasis on reducing the impact of physical illness on the total score. Items are rated on a 4-point severity scale. The HADS produces two scales, one for anxiety (HADS-A) and one for depression (HADS-D), differentiating the two states. Scores of greater than or equal to 11 on either scale indicate a definitive case
Hospital length of stay | up to 45 days
  Time from admission to the hospital to discharge form the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Lomonosov Moscow State University Medical Research and Educational Center, Moscow, Moscow Oblast, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: After publishing
Access Criteria: any application for access the data will be evaluated by ethical commite of LOMONOSOV MOSCOW STATE UNIVERSITY MEDICAL RESEARCH AND EDUCATIONAL CENTER